CLINICAL TRIAL: NCT00344695
Title: Bupropion Treatment for Youth Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3R01CA077081-04S1 (NIH)
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: bupropion SR

SUMMARY:
The purpose of this study is to 1) evaluate the safety and efficacy of two doses of bupropion SR (150mg/day and 300mg/day) when compared to placebo, as an aid to smoking cessation in adolescents and 2) to examine which factors, such as medication adherence, nicotine dependence, and motivation to quit, affect treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 17 years of age
* Smoked at least 6 cigarettes per day
* Exhaled CO greater than or equal to 10 ppm
* Made at least two previous quit attempts
* Weighed at least 90 pounds
* Able to read English at least the 6th grade level
* Motivated to quit smoking as evidenced by willingness to commit to study protocol requirements for the duration of the study
* provided active parental consent and youth assent

Exclusion Criteria:

* Current use of tobacco products other than cigarettes, unless willing to abstain from these products for the study duration
* Current use of other treatments for smoking cessation
* History or current diagnosis of panic disorder, psychosis, bipolar disorder, or eating disorder
* History of abuse or dependence on alcohol or other recreational or prescription drugs in the three months preceding the study
* Current evidence of clinical depression or Attention Deficit/Hyperactivity Disorder
* Use of any psychoactive drug and/or any type of antidepressant with in four weeks of the treatment phase of the study
* Predisposition to seizure or tic disorders or a personal history of a seizure disorder, family history of seizure disorders, or treatment with medication or therapies that increase the risk of seizures
* Significant history of or current clinical evidence of cardiovascular disease
* (Females)Pregnancy (urine pregnancy test), lactation or, if sexually active, unwillingness to use a medically acceptable form of contraception for the duration of the study
* Only one member of a household was allowed to participate in the study concurrently.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Study Completion 2003-04

PRIMARY OUTCOMES:
Biochemically verified 7 day point prevalence abstinence from smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Myra L. Muramoto, MD MPH, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Muramoto ML, Leischow SJ, Sherrill D, Matthews E, Strayer LJ. Randomized, double-blind, placebo-controlled trial of 2 dosages of sustained-release bupropion for adolescent smoking cessation. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1068-74. doi: 10.1001/archpedi.161.11.1068. PMID 17984409